CLINICAL TRIAL: NCT02236533
Title: Healthy Effects of an Innovative Probiotic Pasta
Acronym: SFLABPASTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Parma (Other)
Collaborators: Universita di Verona (Other)
Responsible Party: Principal Investigator, Nicoletta Pellegrini, PhD, Associate Professor, University of Parma
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: SFLAB14
Record Dates: First submitted 2014-07-26; First posted 2014-09-10 (Estimated); Last update posted 2018-11-01 (Actual); Status verified 2018-10

CONDITIONS: OBESITY; INFLAMMATION; DYSLIPIDEMIA; CONSTIPATION
MeSH Terms: conditions — Obesity; Inflammation; Dyslipidemias; Constipation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control pasta (Placebo Comparator): Volunteers were fed with control pasta, without B-glucans and spores of B. coagulans once a day for 12 weeks.
  Interventions: Dietary Supplement: whole grain pasta
- Probiotic Whole Grain Pasta (Experimental): Volunteers were fed with probiotic fortified pasta, including B-glucans and spores of B. coagulans once a day for 12 weeks.
  Interventions: Dietary Supplement: whole grain pasta

INTERVENTIONS:
Dietary Supplement: whole grain pasta — Volunteers were fed with probiotic fortified pasta or control pasta once a day for 12 weeks.

SUMMARY:
The aim of the project was the evaluation of the antioxidant and anti-inflammatory effects of a whole grain pasta, enriched in barley β-glucans and fortified with strains of Bacillus coagulans, versus a control wheat pasta on healthy volunteers, using a parallel randomized controlled trial.

DETAILED DESCRIPTION:
Epidemiological evidences indicate that consumption of whole grains products is associated to a decreased risk for common chronic diseases, as cardiovascular diseases, diabetes, obesity, hypertension and metabolic syndrome. In the present study a whole grain pasta was supplemented with prebiotics and probiotics 'ad hoc' formulated. In detail, pasta was industrially developed after the identification of particular cultivars of wheat and barley, rich in carotenoids, β-glucans (2.6 g/100g pasta), not soluble fibers and antioxidants. Further, pasta was supplemented with spores of Bacillus coagulans, a putative probiotic microorganism, belonging to Lactobacillus family. It is well demonstrated the ability of this microorganism to survive to technological processes and to upper gastro-intesinal tract, in order to exert beneficial effects in the lower gut, as anti-microbial activity, increasing immunological defences as well as improvements in intestinal regularity. Conversely, the control pasta was made from the same cultivar of grain and by the same technological process, but without any supplementation.

In this parallel randomized controlled one arm trial, 40 healthy volunteers were randomly allocated for the consumption of the two kind of pasta once a day, for 12 weeks. At the beginning of the study and every 4 weeks, subjects were asked to provide blood, urine and feces for the evaluation of:

* blood inflammation markers;
* blood lipid and carbohydrate profile;
* blood and urine markers of cardiovascular risk;
* feces profile of microbiota and detection of markers for the healthiness of the gut.

In addition, volunteers filled in different questionnaires regarding their dietary habits, the physical activity and the gut healthiness.

ELIGIBILITY:
Inclusion Criteria:

* Overweight / Obesity
* Lower consumers of fruit and vegetables

Exclusion Criteria:

* Antibiotic treatment within 3 months prior the pasta feeding
* Chronic diseases
* Surgeries
* Consumer of whole grain products
* Dieting
* Pregnant or lactating

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-03; Primary Completion 2014-09 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Variation of plasma lipids | 12 weeks
  Measure of plasma concentrations (mg/dL) of Total-, LDL-, and HDL-Cholesterol; Measure of plasma concentrations (µg/mL) of Non Esterified Fatty Acids (NEFA), Esterified Fatty Acids (EFA) and Short Chain Fatty Acids (SCFA).
  Statistical analysis of the primary outcome was performed within and between each single intervention-arm. Further, a post-hoc subdivision of the study participants by means of a BMI or glycaemia cut-off value was applied, and statistical differences of the primary outcome have been considered.
Variation of fecal microbiota composition | 12 weeks
  By FISH (colony-forming unit, CFU/g).
  Statistical analysis of the primary outcome was performed within and between each single intervention-arm. Further, a post-hoc subdivision of the study participants by means of a BMI or glycaemia cut-off value was applied, and statistical differences of the primary outcome have been considered.
Variation of antioxidant activity on fecal waters | 12 weeks
  Measure of fecal waters FRAP (µmol/L) and TEAC (µmol/L) concentrations.
  Statistical analysis of the primary outcome was performed within and between each single intervention-arm. Further, a post-hoc subdivision of the study participants by means of a BMI or glycaemia cut-off value was applied, and statistical differences of the primary outcome have been considered.

SECONDARY OUTCOMES:
Variation of body weight | 12 weeks
  Measure of body weight (kg).
Variation of serum inflammatory marker concentration | 12 weeks
  Measure of serum IL-2, IL-4, IL-5, IL-6, IL-10, IL-12, IFN-γ,TNF-α, PAI-1, Ghrelin, Leptin, Visfatin, Resistin concentrations (pg/mL).
  Statistical analysis of the secondary outcome was performed within and between each single intervention-arm. Further, a post-hoc subdivision of the study participants by means of a BMI or glycaemia cut-off value was applied, and statistical differences of the secondary outcome have been considered.
Variation of blood pressure | 12 weeks
  Measure of blood pressure (mmHg).
  Statistical analysis of the secondary outcome was performed within and between each single intervention-arm. Further, a post-hoc subdivision of the study participants by means of a BMI or glycaemia cut-off value was applied, and statistical differences of the secondary outcome have been considered.
Variation of body circumferences | 12 weeks
  Measure of waist and hip circumferences (mm).
  Statistical analysis of the secondary outcome was performed within and between each single intervention-arm. Further, a post-hoc subdivision of the study participants by means of a BMI or glycaemia cut-off value was applied, and statistical differences of the secondary outcome have been considered.
Variation of urine antioxidant marker | 12 weeks
  Measurement of betaine in urine (mmol/L).
  Statistical analysis of the secondary outcome was performed within and between each single intervention-arm. Further, a post-hoc subdivision of the study participants by means of a BMI or glycaemia cut-off value was applied, and statistical differences of the secondary outcome have been considered.

CONTACTS AND LOCATIONS:
Overall Officials: Nicoletta Pellegrini, Professor, Principal Investigator — University of Parma
Locations (2):
- Italy (2):
  - University of Parma - Department of Food Sciences, Parma, PR
  - University of Parma, Parma

REFERENCES:
- [Background] Andersson A, Tengblad S, Karlstrom B, Kamal-Eldin A, Landberg R, Basu S, Aman P, Vessby B. Whole-grain foods do not affect insulin sensitivity or markers of lipid peroxidation and inflammation in healthy, moderately overweight subjects. J Nutr. 2007 Jun;137(6):1401-7. doi: 10.1093/jn/137.6.1401. PMID 17513398
- [Background] Behall KM, Scholfield DJ, Hallfrisch J. Diets containing barley significantly reduce lipids in mildly hypercholesterolemic men and women. Am J Clin Nutr. 2004 Nov;80(5):1185-93. doi: 10.1093/ajcn/80.5.1185. PMID 15531664
- [Background] Behall KM, Scholfield DJ, Hallfrisch J. Whole-grain diets reduce blood pressure in mildly hypercholesterolemic men and women. J Am Diet Assoc. 2006 Sep;106(9):1445-9. doi: 10.1016/j.jada.2006.06.010. PMID 16963350
- [Background] Bird AR, Vuaran MS, King RA, Noakes M, Keogh J, Morell MK, Topping DL. Wholegrain foods made from a novel high-amylose barley variety (Himalaya 292) improve indices of bowel health in human subjects. Br J Nutr. 2008 May;99(5):1032-40. doi: 10.1017/S000711450783902X. Epub 2007 Oct 8. PMID 17919346
- [Background] Brouns F, Hemery Y, Price R, Anson NM. Wheat aleurone: separation, composition, health aspects, and potential food use. Crit Rev Food Sci Nutr. 2012;52(6):553-68. doi: 10.1080/10408398.2011.589540. PMID 22452734
- [Background] Brownlee IA, Moore C, Chatfield M, Richardson DP, Ashby P, Kuznesof SA, Jebb SA, Seal CJ. Markers of cardiovascular risk are not changed by increased whole-grain intake: the WHOLEheart study, a randomised, controlled dietary intervention. Br J Nutr. 2010 Jul;104(1):125-34. doi: 10.1017/S0007114510000644. Epub 2010 Mar 23. PMID 20307353
- [Background] Costabile A, Klinder A, Fava F, Napolitano A, Fogliano V, Leonard C, Gibson GR, Tuohy KM. Whole-grain wheat breakfast cereal has a prebiotic effect on the human gut microbiota: a double-blind, placebo-controlled, crossover study. Br J Nutr. 2008 Jan;99(1):110-20. doi: 10.1017/S0007114507793923. Epub 2007 Aug 29. PMID 17761020
- [Background] de Munter JS, Hu FB, Spiegelman D, Franz M, van Dam RM. Whole grain, bran, and germ intake and risk of type 2 diabetes: a prospective cohort study and systematic review. PLoS Med. 2007 Aug;4(8):e261. doi: 10.1371/journal.pmed.0040261. PMID 17760498
- [Background] Dolin BJ. Effects of a proprietary Bacillus coagulans preparation on symptoms of diarrhea-predominant irritable bowel syndrome. Methods Find Exp Clin Pharmacol. 2009 Dec;31(10):655-9. doi: 10.1358/mf.2009.31.10.1441078. PMID 20140275
- [Background] Endres JR, Clewell A, Jade KA, Farber T, Hauswirth J, Schauss AG. Safety assessment of a proprietary preparation of a novel Probiotic, Bacillus coagulans, as a food ingredient. Food Chem Toxicol. 2009 Jun;47(6):1231-8. doi: 10.1016/j.fct.2009.02.018. Epub 2009 Feb 25. PMID 19248815
- [Background] Endres JR, Qureshi I, Farber T, Hauswirth J, Hirka G, Pasics I, Schauss AG. One-year chronic oral toxicity with combined reproduction toxicity study of a novel probiotic, Bacillus coagulans, as a food ingredient. Food Chem Toxicol. 2011 May;49(5):1174-82. doi: 10.1016/j.fct.2011.02.012. Epub 2011 Feb 19. PMID 21338652
- [Background] Grasten SM, Juntunen KS, Poutanen KS, Gylling HK, Miettinen TA, Mykkanen HM. Rye bread improves bowel function and decreases the concentrations of some compounds that are putative colon cancer risk markers in middle-aged women and men. J Nutr. 2000 Sep;130(9):2215-21. doi: 10.1093/jn/130.9.2215. PMID 10958815
- [Background] Honda H, Gibson GR, Farmer S, Keller D, McCartney AL. Use of a continuous culture fermentation system to investigate the effect of GanedenBC30 (Bacillus coagulans GBI-30, 6086) supplementation on pathogen survival in the human gut microbiota. Anaerobe. 2011 Feb;17(1):36-42. doi: 10.1016/j.anaerobe.2010.12.006. Epub 2010 Dec 30. PMID 21195203
- [Background] Hun L. Bacillus coagulans significantly improved abdominal pain and bloating in patients with IBS. Postgrad Med. 2009 Mar;121(2):119-24. doi: 10.3810/pgm.2009.03.1984. PMID 19332970
- [Background] Kalman DS, Schwartz HI, Alvarez P, Feldman S, Pezzullo JC, Krieger DR. A prospective, randomized, double-blind, placebo-controlled parallel-group dual site trial to evaluate the effects of a Bacillus coagulans-based product on functional intestinal gas symptoms. BMC Gastroenterol. 2009 Nov 18;9:85. doi: 10.1186/1471-230X-9-85. PMID 19922649
- [Background] Katcher HI, Legro RS, Kunselman AR, Gillies PJ, Demers LM, Bagshaw DM, Kris-Etherton PM. The effects of a whole grain-enriched hypocaloric diet on cardiovascular disease risk factors in men and women with metabolic syndrome. Am J Clin Nutr. 2008 Jan;87(1):79-90. doi: 10.1093/ajcn/87.1.79. PMID 18175740
- [Background] Kimmel M, Keller D, Farmer S, Warrino DE. A controlled clinical trial to evaluate the effect of GanedenBC(30) on immunological markers. Methods Find Exp Clin Pharmacol. 2010 Mar;32(2):129-32. doi: 10.1358/mf.2010.32.2.1423881. PMID 20401350
- [Background] Lappi J, Kolehmainen M, Mykkanen H, Poutanen K. Do large intestinal events explain the protective effects of whole grain foods against type 2 diabetes? Crit Rev Food Sci Nutr. 2013;53(6):631-40. doi: 10.1080/10408398.2010.550388. PMID 23627504
- [Background] Lappi J, Salojarvi J, Kolehmainen M, Mykkanen H, Poutanen K, de Vos WM, Salonen A. Intake of whole-grain and fiber-rich rye bread versus refined wheat bread does not differentiate intestinal microbiota composition in Finnish adults with metabolic syndrome. J Nutr. 2013 May;143(5):648-55. doi: 10.3945/jn.112.172668. Epub 2013 Mar 20. PMID 23514765
- [Background] Larsson SC, Giovannucci E, Bergkvist L, Wolk A. Whole grain consumption and risk of colorectal cancer: a population-based cohort of 60,000 women. Br J Cancer. 2005 May 9;92(9):1803-7. doi: 10.1038/sj.bjc.6602543. PMID 15827552
- [Background] Leinonen KS, Poutanen KS, Mykkanen HM. Rye bread decreases serum total and LDL cholesterol in men with moderately elevated serum cholesterol. J Nutr. 2000 Feb;130(2):164-70. doi: 10.1093/jn/130.2.164. PMID 10720164
- [Background] Mandel DR, Eichas K, Holmes J. Bacillus coagulans: a viable adjunct therapy for relieving symptoms of rheumatoid arthritis according to a randomized, controlled trial. BMC Complement Altern Med. 2010 Jan 12;10:1. doi: 10.1186/1472-6882-10-1. PMID 20067641
- [Background] Martinez I, Lattimer JM, Hubach KL, Case JA, Yang J, Weber CG, Louk JA, Rose DJ, Kyureghian G, Peterson DA, Haub MD, Walter J. Gut microbiome composition is linked to whole grain-induced immunological improvements. ISME J. 2013 Feb;7(2):269-80. doi: 10.1038/ismej.2012.104. Epub 2012 Oct 4. PMID 23038174
- [Background] McIntosh GH, Noakes M, Royle PJ, Foster PR. Whole-grain rye and wheat foods and markers of bowel health in overweight middle-aged men. Am J Clin Nutr. 2003 Apr;77(4):967-74. doi: 10.1093/ajcn/77.4.967. PMID 12663299
- [Background] Mellen PB, Walsh TF, Herrington DM. Whole grain intake and cardiovascular disease: a meta-analysis. Nutr Metab Cardiovasc Dis. 2008 May;18(4):283-90. doi: 10.1016/j.numecd.2006.12.008. Epub 2007 Apr 20. PMID 17449231
- [Background] Nilsson AC, Ostman EM, Holst JJ, Bjorck IM. Including indigestible carbohydrates in the evening meal of healthy subjects improves glucose tolerance, lowers inflammatory markers, and increases satiety after a subsequent standardized breakfast. J Nutr. 2008 Apr;138(4):732-9. doi: 10.1093/jn/138.4.732. PMID 18356328
- [Background] Pellegrini N, Del Rio D, Colombi B, Bianchi M, Brighenti F. Application of the 2,2'-azinobis(3-ethylbenzothiazoline-6-sulfonic acid) radical cation assay to a flow injection system for the evaluation of antioxidant activity of some pure compounds and beverages. J Agric Food Chem. 2003 Jan 1;51(1):260-4. doi: 10.1021/jf020657z. PMID 12502418
- [Background] Pereira MA, Jacobs DR Jr, Pins JJ, Raatz SK, Gross MD, Slavin JL, Seaquist ER. Effect of whole grains on insulin sensitivity in overweight hyperinsulinemic adults. Am J Clin Nutr. 2002 May;75(5):848-55. doi: 10.1093/ajcn/75.5.848. PMID 11976158
- [Background] Priebe MG, Wang H, Weening D, Schepers M, Preston T, Vonk RJ. Factors related to colonic fermentation of nondigestible carbohydrates of a previous evening meal increase tissue glucose uptake and moderate glucose-associated inflammation. Am J Clin Nutr. 2010 Jan;91(1):90-7. doi: 10.3945/ajcn.2009.28521. Epub 2009 Nov 4. PMID 19889821
- [Background] Ross AB, Bruce SJ, Blondel-Lubrano A, Oguey-Araymon S, Beaumont M, Bourgeois A, Nielsen-Moennoz C, Vigo M, Fay LB, Kochhar S, Bibiloni R, Pittet AC, Emady-Azar S, Grathwohl D, Rezzi S. A whole-grain cereal-rich diet increases plasma betaine, and tends to decrease total and LDL-cholesterol compared with a refined-grain diet in healthy subjects. Br J Nutr. 2011 May;105(10):1492-502. doi: 10.1017/S0007114510005209. Epub 2011 Jan 28. PMID 21272402
- [Background] Sahyoun NR, Jacques PF, Zhang XL, Juan W, McKeown NM. Whole-grain intake is inversely associated with the metabolic syndrome and mortality in older adults. Am J Clin Nutr. 2006 Jan;83(1):124-31. doi: 10.1093/ajcn/83.1.124. PMID 16400060
- [Background] Scazzina F, Siebenhandl-Ehn S, Pellegrini N. The effect of dietary fibre on reducing the glycaemic index of bread. Br J Nutr. 2013 Apr 14;109(7):1163-74. doi: 10.1017/S0007114513000032. Epub 2013 Feb 18. PMID 23414580
- [Background] Emerick RE. The politics of psychiatric self-help: political factions, interactional support, and group longevity in a social movement. Soc Sci Med. 1991;32(10):1121-8. doi: 10.1016/0277-9536(91)90088-t. PMID 2068595
- [Background] Valtuena S, Pellegrini N, Franzini L, Bianchi MA, Ardigo D, Del Rio D, Piatti P, Scazzina F, Zavaroni I, Brighenti F. Food selection based on total antioxidant capacity can modify antioxidant intake, systemic inflammation, and liver function without altering markers of oxidative stress. Am J Clin Nutr. 2008 May;87(5):1290-7. doi: 10.1093/ajcn/87.5.1290. PMID 18469252
- [Background] Whelton SP, Hyre AD, Pedersen B, Yi Y, Whelton PK, He J. Effect of dietary fiber intake on blood pressure: a meta-analysis of randomized, controlled clinical trials. J Hypertens. 2005 Mar;23(3):475-81. doi: 10.1097/01.hjh.0000160199.51158.cf. PMID 15716684
- [Background] Ye EQ, Chacko SA, Chou EL, Kugizaki M, Liu S. Greater whole-grain intake is associated with lower risk of type 2 diabetes, cardiovascular disease, and weight gain. J Nutr. 2012 Jul;142(7):1304-13. doi: 10.3945/jn.111.155325. Epub 2012 May 30. PMID 22649266
- [Derived] Angelino D, Martina A, Rosi A, Veronesi L, Antonini M, Mennella I, Vitaglione P, Grioni S, Brighenti F, Zavaroni I, Fares C, Torriani S, Pellegrini N. Glucose- and Lipid-Related Biomarkers Are Affected in Healthy Obese or Hyperglycemic Adults Consuming a Whole-Grain Pasta Enriched in Prebiotics and Probiotics: A 12-Week Randomized Controlled Trial. J Nutr. 2019 Oct 1;149(10):1714-1723. doi: 10.1093/jn/nxz071. PMID 31162597